CLINICAL TRIAL: NCT00962338
Title: Pain and Convalescence After Laparoscopic Groin Hernia Repair
Acronym: Lap-Lyske
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Mette Astrup Madsen, M.D., Zealand University Hospital
Other Study IDs: SJ-125
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Inguinal Hernia; Convalescence
Keywords: convalescence; pain; nausea; vomiting; sexual dysfunction
MeSH Terms: conditions — Hernia, Inguinal; Convalescence; Pain; Nausea; Vomiting; Sexual Dysfunction, Physiological | interventions — tetra-4-amidinophenoxypropane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- lap. inguinal herniorrhaphy: Patients undergoing planned lap. inguinal herniorrhaphy
  Interventions: Behavioral: Information

INTERVENTIONS:
Behavioral: Information — Information on short convalescence (1 day). Example: Operated today and getting started with normal activities again tomorrow.
  Other Names: Groin hernia repair; TAPP; Convalescence

SUMMARY:
The investigators want to identify limiting factors for short convalescence after laparoscopic groin hernia repair. Before the operation patients are given intensive structured information about one day´s convalescence. Patients fill out questionnaire before operation about several clinically relevant parameters. This is also done first 3 days after operation and after 1 month and 6 months. The patients are seen for clinical control at 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* planned laparoscopic inguinal or femoral herniorrhaphy
* ASA class I-II
* speak and read danish

Exclusion Criteria:

* converting to open operation
* low compliance (dementia, psychiatric disorder)
* use of morphine or similar drugs daily in the last month
* complications to the operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population are from Region Sjaelland and are planned for laparoscopic inguinal or femoral herniorrhaphy. Single university hospital department i Denmark.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
duration of convalescence | 3 weeks in average

SECONDARY OUTCOMES:
Pain scores on visual analog scale and verbal rating scale | 6 months
  daily first 4 days, after 1 and 6 months
fatigue scores on numeric rating scale (1-10) | 6 months
  daily first 4 days, 1 and 6 months
sexual dysfunction | 6 months
nausea scores on verbal rating scale | 3 days
vomiting | 3 days
wellbeing scores on visual analog scale | 6 months
Hospital anxiety and depression scale (HAD) | Baseline (before operation)
Pain catastrophizing scale (PCS) | Baseline (before operation)
Activity assessment scale (AAS) | Baseline (before operation)
  Functional status

CONTACTS AND LOCATIONS:
Overall Officials: Mette A Tolver, M.D., Principal Investigator — University Hospital Køge
Locations (1):
- University Hospital Køge, Koege, Region Sjælland, Denmark

REFERENCES:
- [Derived] Tolver MA, Rosenberg J. Pain during sexual activity before and after laparoscopic inguinal hernia repair. Surg Endosc. 2015 Dec;29(12):3722-5. doi: 10.1007/s00464-015-4143-8. Epub 2015 Mar 18. PMID 25783834
- [Derived] Tolver MA, Strandfelt P, Rosenberg J, Bisgaard T. Female gender is a risk factor for pain, discomfort, and fatigue after laparoscopic groin hernia repair. Hernia. 2013 Jun;17(3):321-7. doi: 10.1007/s10029-012-0956-8. Epub 2012 Jul 12. PMID 22790511